CLINICAL TRIAL: NCT01339351
Title: Teleconference Group: Breast Cancer in African Americans
Brief Title: Teleconference Group: Breast Cancer in African Americans (STORY)
Acronym: STORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Sue Heiney, Research Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2004-62
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; social connection
MeSH Terms: conditions — Breast Neoplasms | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Psychosocial Care (No Intervention): Participants are free to use any psychosocial care available to cancer patients. No restrictions to participation in other groups or services.
- Therapeutic Group by teleconference (Experimental): ten 90 minute group sessions by teleconference. Lead by social workers. Sessions focus on information, story sharing and coping.
  Interventions: Behavioral: Therapeutic Group by Teleconference

INTERVENTIONS:
Behavioral: Therapeutic Group by Teleconference — 10 sessions
  Other Names: Support group
  Arms: Therapeutic Group by teleconference

SUMMARY:
African American women with breast cancer have decreased quality of life (and mood when compared to European American. Research has not examined the effectiveness of therapeutic group for African American women with breast cancer even though positive effects are well established for Caucasians. The aims of the randomized clinical trial are to determine the effectiveness of TG by teleconference for African American women with breast cancer and what factors may impact on the intervention. The primary hypothesis is that participants in the intervention group will have significantly greater cancer knowledge, less fear, less isolation, better social connection, better mood, and better QOL when compared to a control group receiving usual psychosocial care. Two hundred forty African American women with breast cancer will be recruited. Intervention participants attend eight weekly 90 minute sessions by teleconference and two follow-up boosters. Each culturally appropriate session contains the story, information and group processes of connection, commonality and catharsis. Information focuses on increasing self care and stress management knowledge while countering myths and taboos. Story capitalizes on African American oral traditions by discussing coping parables. Group processes provide an alternative source of social support and opportunities to express feelings. Control group subjects receive standard psychosocial care (the use of any support programs or services locally or nationally. Testing will occur at baseline, after 10 group sessions and 16 weeks post baseline. The study findings are expected to inform about the effectiveness of therapeutic groups in African American women with breast cancer and lay the groundwork for exploring if reducing disparities in psychosocial care have a health benefit.

DETAILED DESCRIPTION:
A. Specific Aims Aim One The major aim of the proposed study is to compare the effects of a TG by conference call for AAWBC with usual psychosocial care. We hypothesize that AAWBC who receive the TG by teleconference will have significantly greater cancer knowledge, less fear, less isolation, better social connection, better mood, and better QOL than a control group receiving usual psychosocial care.

Aim One A: Substantiate intervention integrity (purity, dosage, specificity and interventionist competency) of first 14 waves of study.

Aim One B: Establish reliability and validity of measures (Profile of Mood States and Functional Assessment of Cancer Therapy - Breast Cancer Version, Social Support Questionnaire) Aim Two To have a strong intervention, it is essential to identify the processes of change that lead to beneficial outcomes.29, 30 Therefore, the second aim of the proposed study is to identify the mediators of the intervention that predict successful treatment outcomes.

Aim Three Since it is particularly important to identify AA women's characteristics and sociocultural factors which may affect their responses to the intervention,30, 31 the third aim of the study is to identify the effects of demographic, health and socio-cultural variables as moderators of treatment effects on social connection, and QOL.

Aim Three A: Examine baseline moderators and concept of social connection to establish associations.

C. EXPERIMENTAL DESIGN & METHODS Design The proposed study will be conducted as a multiple-group randomized trial to compare the TG intervention with a control group receiving usual psychosocial care. A maximum of 10 subjects will be assigned randomly to each of two groups during a common time period, with one group receiving the TG intervention and the other receiving usual care. The randomization will be stratified by treatment type (chemo therapy only or radiation therapy only or chemotherapy and radiation therapy combined). Multiple time periods will be used to achieve the required number of subjects for the entire trial. Subjects will be evaluated at three time points in a repeated measures fashion: (1) at baseline before the intervention begins, (2) at the end of the intervention period, and (3) 16 weeks from baseline. Mediating, moderating and outcome variable data will be collected at all three time periods.

These measurement times have been chosen for several reasons. The intervention will be delivered during the stressful time after diagnosis when the patient is facing fears, side effects (especially body image changes), and negative community attitudes. During this time, patients are challenged to learn about the disease and its treatment and are emotionally open to using positive coping strategies.133-136 The T-2 measurement will provide information on the immediate effects of the treatment and T-3 will provide information on the sustainability of the intervention effects.

Setting South Carolina is an ideal setting within which to test the proposed intervention, TG by teleconference. AA represent about 31 % of the population. Unlike other parts of the US, SC is mostly rural (and 46 % of its AA are rural) and the AA population has experienced very little in-migration over the past several centuries.137 Furthermore, religious affiliation is largely fundamentalist Christian (African Methodist Episcopal, Baptist and Pentecostal Churches),138 and a spiritual focus permeates the community, which is known as the "Buckle" of the Bible Belt.

Major statewide initiatives to decrease health disparities are in progress and these efforts have resulted in multiple networks for communication with key SC community leaders and health providers. We will use the Cancer Research Network, SC Cancer Alliance, Women's Cancer Coalition and the Best Chance Network to enhance recruitment efforts.

Palmetto Health and the University of South Carolina are exceptional bases from which to conduct this research. Palmetto Health is South Carolina's most comprehensive health resource, a locally owned, not-for-profit healthcare system with Palmetto Health Baptist Easley in upstate SC and two Columbia hospitals, Palmetto Health Baptist and Palmetto Health Richland. Palmetto Health's Comprehensive Breast Center (PHCBC) was established to improve treatment using national guidelines and decrease mortality. Over the past several years, major strides have been made in attaining these goals through detection of smaller tumors and use of sentinel node biopsy. Two multi-disciplinary and multi-specialty breast cancer tumor conferences are held weekly. Additionally, Palmetto Health has made a strong commitment to decrease health disparities in the communities it serves through its Cancer Community Health Initiative. The 6 year-old initiative has targeted AAs and is working to improve individual and community health by providing services to underserved and uninsured populations especially cancer screening.

One of the oldest and most comprehensive public universities in the United States, USC has been designated a research institution of "very high research activity," the only university in South Carolina to have this designation, granted to 62 public and 32 private research institutions. University libraries in Columbia house over 7,000,000 processed items including 2,639,171 volumes and approximately 4,075,413 units in microform. Some 17,405 current periodicals are received. Thomas Cooper Library. Included in the seating are more than 900 private locked facilities for faculty and graduate students involved in research. Special areas in the library include the Student Computer Labs, the Science Library, Special Collections, and the Map Library. Access to the collection is obtained through the USCAN/NOTIS Online Card Catalog with terminals located throughout the building. CD ROM stations are available for user searching of multiple databases. The Thomas Cooper Library offers access to literature from international sources through the on-line computer-assisted reference department. The computerized reference service provides bibliographic citations, statistics, and international news from recent literature on a wide range of subjects. This service is particularly strong in the natural and social sciences. Also included are government activities, publications, and grant sources. Data bases in nursing include Medline, Nursing and Allied Health, and Health Planning and Administration. Data bases related to nursing include Psychological Abstracts and Mental Health Abstracts. New data bases are added regularly, and information on them is available in the Reference Department.

The majority of participants in the proposed study will be recruited from the two cancer treatment sites within Palmetto Health, which treats about 600 breast cancer patients annually. Of those, more than 225 are AAWBC. Other recruitment will be statewide.

ELIGIBILITY:
Inclusion Criteria:

* US born
* African American women
* age 21 or older
* diagnosed with invasive/infiltrating ductal carcinoma
* reside in South Carolina or the borders of North Carolina or Georgia

Exclusion Criteria:

* Non-english speaking
* diagnosed with metastatic disease at diagnosis
* have a major cognitive impairment
* have a current diagnosis of psychosis
* are undergoing concurrent treatment for another form of cancer (except basal cell or squamous cell of skin)
* Participation in another behavioral trial

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2005-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Social connection | Participants are assessed at time one (baseline/pretest) and followed for 16 weeks
  Measured using the social well-being scale from the FACT-B

SECONDARY OUTCOMES:
Fatalism | Participants are assessed at time one (baseline/pretest) and followed for 16 weeks
  Powe Fatalism Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sue P. Heiney, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Result] Heiney SP, Adams SA, Wells LM, Johnson H. Evaluation of conceptual framework for recruitment of African American patients with breast cancer. Oncol Nurs Forum. 2010 May;37(3):E160-7. doi: 10.1188/10.ONF.E160-E167. PMID 20439201